CLINICAL TRIAL: NCT03172195
Title: Detection of Herpesvirus DNA (CMV, EBV, HHV-6 and HSV) in Colonic Tissue: Impact on Ulcerative Colitis Flare-up
Acronym: VIRCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: * Lack of inclusion
  * Inability to open investigator centers due to lack of budget
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1708033; ANSM (Other: 2017-A00988-45)
Record Dates: First submitted 2017-05-23; First posted 2017-06-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Colitis, Ulcerative
Keywords: ulcerative colitis; inflammation; immunosuppressive drugs; herpesvirus; qPCR; colonic mucosa
MeSH Terms: conditions — Colitis, Ulcerative; Inflammation; Herpes Simplex | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with ulcerative colitis (Experimental): Patients with ulcerative colitis will have a rectosigmoidoscopy, biopsies and blood sample.
  Interventions: Procedure: rectosigmoidoscopy; Biological: biopsies; Biological: blood sample

INTERVENTIONS:
Procedure: rectosigmoidoscopy — A rectosigmoidoscopy will be realized and two fragments will be collected.
Biological: biopsies — For this study, two biopsies in healthy area and two biopsies in ulcer will be collected.
Biological: blood sample — Blood sample will be collected in more.

SUMMARY:
Flare-up of ulcerative colitis (UC) is characterized by the inflammation of colon mucosa that requires the use of immunosuppressive therapies. In previous studies, the active role of cytomegalovirus (CMV) has been demonstrated, with a correlation between the cytomegalovirus DNA ((deoxyribonucleic acid) load in the inflamed tissue and the resistance to successive lines of immunosuppressive therapy (Roblin et al., Am J Gastroenterol 2011). The main aim of this monocentric prospective study is to evaluate the DNA viral load by qPCR (Polymerase Chain Reaction) of 3 herpesviruses (Epstein-Barr virus, herpes virus 6 and herpes simplex) together with that of CMV in colonic mucosa depending of the local inflammation (endoscopically normal region, inflamed mucosa or ulcer) in patients suffering of moderate to severe UC flare-up (Mayo score >6 with endoscopic score higher or equal than 2). The viral load will also be correlated to the Mayo endoscopic score and the response to immunosuppressive drugs (steroid and anti-TNF (Tumor Necrosis Factor) monoclonal antibodies).

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Voluntary to participate to the study
* Flare-up of ulcerative colitis with Mayo score >6
* Ability to receive steroid or anti-TNF therapy
* Agree the rectosigmoidoscopy and the therapies

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Disagree the rectosigmoidoscopy or the therapies
* Participation to the evaluation of a new therapy
* Colectomy (partial or total)
* Contraindication of steroid or anti-TNF therapy
* Anticoagulant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with different viral load in the colonic mucosa | day 1
  Different viral loads are a composite outcome : viral load of CMV, EBV, HHV-6 and HSV.
  It will be measured by Polymerase Chain Reaction technical in colonic mucosa

SECONDARY OUTCOMES:
Correlation of the different viral loads with the Mayo endoscopic score | Day 1
  Different viral loads are a composite outcome : viral load of CMV, EBV, HHV-6 and HSV.
  It will be measured by Polymerase Chain Reaction technical in colonic mucosa The Mayo endoscopic score integrate the severity from lesions of colonic mucosa measured by rectosigmoidoscopy
Correlation of the different viral loads with the steroid treatment response | up to 24 months
  Different viral loads are a composite outcome : viral load of CMV, EBV, HHV-6 and HSV.
  It will be measured by Polymerase Chain Reaction technical in colonic mucosa.
  Steroid treatment response is defined by clinic mayo score < 3 measured by rectosigmoidoscopy.
Correlation of the different viral loads with the anti-TNF treatment response | up to 24 months
  Different viral loads are a composite outcome : viral load of CMV, EBV, HHV-6 and HSV.
  It will be measured by Polymerase Chain Reaction technical in colonic mucosa. anti-TNF treatment response is defined by clinic mayo score < 3 measured by rectosigmoidoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Roblin, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No